CLINICAL TRIAL: NCT01109381
Title: A Single-centre, Open-label, Non-controlled, Exploratory Safety and Efficacy Clinical Trial of GT08 in Volunteers and Patients Who Are Infected With Helicobacter Pylori
Brief Title: Safety and Efficacy Study of a Non-antibiotic Treatment for the Eradication of Helicobacter Pylori
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor efficacy (2 of 31 completing participants with H.pylori eradication)
Sponsor: Synergy Pharmaceuticals Pte. Ltd. (Industry)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GT08-01
Record Dates: First submitted 2010-04-20; First posted 2010-04-23 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: bacterial infections; anti-infective agents; gastrointestinal agents; antibacterial agents; omeprazole; lauric acid; n-acetylcysteine; helicobacter infections; helicobacter pylori; non-antibiotic treatment
MeSH Terms: conditions — Bacterial Infections; Helicobacter Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with GT08 (Experimental): Initial phase - omeprazole, N-acetyl cysteine (NAC), lauric acid dose and duration titration from 1 up to 14 days of treatment. Secondary phase - 14 days treatment with omeprazole, NAC, lauric acid
  Interventions: Drug: GT08

INTERVENTIONS:
Drug: GT08 — GT08 is the combination of omeprazole 40mg daily, lauric acid 150-300mg daily, NAC 1.2 - 2g daily

SUMMARY:
At present, triple therapy is recommended by various guidelines for the treatment of Helicobacter pylori (H.pylori) infection. Recent studies have shown increasing resistance of H.pylori to commonly used antibiotics used in triple therapy. This study explores a non-antibiotic treatment regime for H.pylori that uses lauric acid as the primary anti-microbial agent. The study hypothesis is that Lauric acid works synergistically with omeprazole following administration of a mucolytic agent to kill H.pylori topically in the stomach.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent prior to any study procedure
* Age at least 21 years and up to 70 years
* If female of childbearing potential who is sexually active, agrees to use acceptable methods of birth control throughout the study. Acceptable methods of birth control are: hormonal contraceptives (birth control pills), intrauterine device (IUD), diaphragm with spermicide, condom, vasectomy.

Additional Inclusion Criteria for Initial Phase only

* Healthy volunteers - can have gastrointestinal or other symptoms if these do not require medical treatment and are considered by the investigator to be clinically minor and irrelevant to the conduct of the study.
* Positive laboratory serology for H.pylori
* Positive Urea Breath Test for H.pylori
* Willing to undergo two gastroscopy procedures

Additional Inclusion Criteria for Secondary Phase only

* Either healthy volunteers or patients attending gastroenterology outpatient clinic - can have gastrointestinal or other symptoms if these are considered by the investigator to be clinically minor or irrelevant to the conduct of the study.
* Positive diagnosis of current H.pylori infection, as diagnosed by positive Urea Breath Test and at least one of the following: 1) Positive laboratory serology for H.pylori, 2) known positive Campylobacter-like organism (CLO) test or H.pylori culture from a gastroscopy performed in the 1 year prior to Screening.

Exclusion Criteria:

* Pregnant or breast feeding.
* Clinically significant gastric disease, in the opinion of the investigator.
* Significant disease or disorder on general medical examination, in the opinion of the investigator (general, respiratory, cardiovascular, renal, hepatic, neurological, bleeding tendency etc).
* Regular or intermittent use of antibiotics, non-steroidal anti-inflammatory drugs (NSAIDs), anticoagulants or antiplatelet medications is expected during the trial period.
* Cessation of proton pump inhibitor or H2-blocker therapy for 2 weeks prior to Urea Breath Test is likely to not be in the best interests of the participant.
* Laboratory values on blood testing that are outside of the laboratory normal range and considered clinically relevant by the investigator: the following will be screened Haemoglobin (Hb), bilirubin, aspartate transaminase (AST), alanine transaminase (ALT), serum albumin, Alkaline Phosphatase, Urea, sodium (Na), potassium (K), creatinine (CRE).
* Any contraindication to treatment with omeprazole, N-acetyl cysteine (NAC), or sodium bicarbonate.
* Any evidence of organic or psychiatric disorders likely to result in poor compliance in the opinion of the investigator.
* Previous participation in this trial at any time, or participation in any other clinical trial within the previous 3 months.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ling Khoon Lin, MRCP, DPhil, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited, with the first volunteer consenting for screening on 13 May 2010. A total of 205 healthy volunteers were screened for the study, with 164 not being infected with H.pylori and 8 not entering the trial for other inclusion/exclusion reasons.
Pre-assignment Details: No group assignment - all participants included were to receive trial treatment. Following consent to take part in the study, participants had a pre-treatment gastroscopy to exclude significant existing upper GI disease. Then all received omeprazole 40mg daily for 1 week prior to receiving the investigational GT08 treatment.
Groups:
- GT08: Initial phase - omeprazole, N-acetylcysteine (NAC), lauric acid dose and duration titration from 1 up to 14 days of treatment. Secondary phase - 14 days treatment with omeprazole, NAC, lauric acid
  GT08 : omeprazole 40mg daily, lauric acid 150-300mg daily, NAC 1.2 - 2g daily
Period: Overall Study
Arm/Group | GT08
Started | 33
Completed | 31
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Initial phase - omeprazole, NAC, lauric acid dose and duration titration from 1 up to 14 days of treatment. Secondary phase - 14 days treatment with omeprazole, NAC, lauric acid
  GT08 : omeprazole 40mg daily, lauric acid 150-300mg daily, NAC 1.2 - 2g daily
Arm/Group | Treatment
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Region of Enrollment [Number; unit: participants]
  Singapore | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Eradication of H.Pylori Infection
Description: Eradication as measured by negative Urea Breath Test 4-6 weeks following completion of treatment
Time Frame: 4-6 weeks following treatment
Population: Two participants did not complete the study, one discontinuing after experiencing adverse events while receiving only the initial study omeprazole, and the other participant left Singapore before they had their final urea breath test. All other study participants were analysed for efficacy.
Measure: Number; unit: participants
Groups:
- Treatment With GT08: Initial phase - omeprazole, N-acetyl cysteine (NAC), lauric acid dose and duration titration from 1 up to 14 days of treatment. Secondary phase - 14 days treatment with omeprazole, NAC, lauric acid
  GT08 means treatment with omeprazole 40mg daily, lauric acid 150-300mg daily, and NAC 1.2 - 2g daily
Arm/Group | Treatment With GT08
Number analyzed (Participants) | 31
participants | 2

2. Primary Outcome: Absence of Significant Gastric Abnormality Post-treatment (Initial Phase)
Description: Gastroscopy pre- and post-treatment will be performed in the Initial Phase (20 participants), with the goal of excluding significant gastric abnormality at baseline and after treatment (e.g. gastric ulceration arising following the treatment).
Time Frame: up to 14 days of treatment
Population: All 21 Initial Phase participants had a pretreatment gastroscopy, and 20 had post-treatment gastroscopy (one participant prematurely discontinued the study prior to receiving GT08, and the participant later lost to follow up had a post-treatment gastroscopy before being lost to follow up)
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
participants | 20

3. Secondary Outcome: Assessment of Adverse Events (AE)
Description: Adverse event data will be collected in response to neutral questioning.
Time Frame: AE commencing within 30 days of initiation of treatment, followed until resolution
Population: All participants entering the study are included in the safety analysis
Measure: Number; unit: participants
Groups:
- Treatment: Initial phase - omeprazole, NAC (N-acetyl cysteine), lauric acid with dose and duration titration from 1 up to 14 days of treatment. Secondary phase - 14 days treatment with omeprazole, NAC, lauric acid
  GT08 is the combination of omeprazole 40mg daily, lauric acid 150-300mg daily, NAC 1.2 - 2g daily
Arm/Group | Treatment
Number analyzed (Participants) | 33
participants | 12

ADVERSE EVENTS:
Time Frame: From the time of study entry until 30 days after finishing study treatments or until resolution.
Description: Adverse events were recorded by open questioning at study visits, and also recorded if there was any other contact between the participant and the study centre.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 12/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=33)
abdominal pain or discomfort (Gastrointestinal disorders) | 3 (3) — Mild abdominal pain, discomfort or stomach cramps recorded in 3 participants, Severity mild. Resolved within 48 hours, and considered unlikely related to study medication.
flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 7 (7) — Runny nose, cough, upper respiratory tract infection, viral infection or sore throat
nausea or vomiting (Gastrointestinal disorders) | 3 (3) — severity mild, none leading to discontinuation of therapy
joint swelling and pain (Musculoskeletal and connective tissue disorders) | 2 (3) — husband and wife experienced sore throat after completing GT08 therapy, developing mildly sore joints some 3 weeks later. Resolved other than his knee being diagnosed as mild patello-femoral OA with some persistent pain. Unlikely related to GT08.

LIMITATIONS AND CAVEATS:
The trial has no control group. All participants had current H.pylori infection at study entry. Only two participants had this infection eradicated, making an efficacy control group unnecessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less